CLINICAL TRIAL: NCT01226641
Title: Usefulness of a Telemedicine System for OSA Patients Follow-up With High Cardiovascular Risk
Acronym: TELESAS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Initiative Pour la Sante (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: InitiativePS-TELESAS
Record Dates: First submitted 2010-10-20; First posted 2010-10-22 (Estimated); Last update posted 2013-01-17 (Estimated); Status verified 2013-01

CONDITIONS: Sleep Apnea, Obstructive; Obstructive Sleep Apnea Syndrome
Keywords: Obstructive Sleep Apnea Syndrome; SCORE; Telemedicine; Arterial blood pressure; Daily physical activity
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Telemedecine (Experimental): CPAP treatment with telemedicine system
  Interventions: Device: Telemedicine
- Standard Care (Active Comparator): Standard care, including CPAP
  Interventions: Device: Standard care

INTERVENTIONS:
Device: Telemedicine — CPAP treatment with telemedicine system
  Arms: Telemedecine
Device: Standard care — Standard care, including CPAP
  Arms: Standard Care

SUMMARY:
The aim of this study is to determine the usefulness of a telemedicine system for the follow-up of OSA patients with a high cardiovascular risk. Our hypothesis is that the telemedicine system will enhance compliance and thus reduce self-measured blood pressure.

DETAILED DESCRIPTION:
The obstructive sleep apnea syndrome (OSAS) corresponds to repeated epochs of complete or incomplete pharynx collapses occurring during sleep. The Continuous Positive Airway Pressure is the gold standard treatment for OSAS. It consists of air insufflation in upper airways with a pressure of about 5 to 15 cm of water with a facial or nasal mask. CPAP treatment reduces cardiovascular morbi-mortality.

OSAS is associated with cardiovascular mortality. A dose response effect exists between severity and arterial blood pressure. A recent meta-analysis has shown in unselected OSAS patients with or without hypertension, treated or non-treated for hypertension, CPAP reduces 24 h ambulatory blood pressure of approximately 2 mmHg. This decrease corresponds to a significant reduction in cardiovascular risk.

The aim of the present study is to include OSAS patients with a high cardiovascular risk and to measure the effect of CPAP on home measurements of arterial blood pressure. This controlled randomized trial will compare the effect CPAP on arterial blood pressure in a group with a telemedicine system versus a group with standard home care CPAP treatment.

An interim analysis will be carried out when 100 patients have been included in the study.

ELIGIBILITY:
Inclusion Criteria:

* 18 to 85 years old men and women
* stable patient
* BMI<40kg/m²
* OSA patients diagnosed with polysomnography or polygraphy
* SCORE>5% and/or cardiovascular disease pas history :
* transient ischemic attack, stroke, cerebral haemorrhagy
* myocardial infraction, angor, coronary revascularization, arteriopathy, aortic aneurism

Exclusion Criteria:

* central sleep apnea syndrome
* SCORE<5%
* cardiac failure
* past history of hypercapnic chronic respiratory failure
* past history of severe or intercurrent pathology which can not allow the patient follow-up
* Incapacitated patients in accordance with article L 1121-6 of the public health code
* patients taking part in another clinical trial

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 107 (Actual)
Dates: Start 2009-07; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Home Arterial Blood Pressure | Home arterial Blood Pressure is assessed at week 1
  the primary outcome is assessed at weeks 1 and 16 for the both groups, moreover home arterial blood pressure is assessed each day, 2 times : morning and afternoon in the telemedicine group.
Home Arterial Blood Pressure | Home arterial Blood Pressure is assessed at week 16
  the primary outcome is assessed at weeks 1 and 16 for the both groups, moreover home arterial blood pressure is assessed each day, 2 times : morning and afternoon in the telemedicine group.

SECONDARY OUTCOMES:
CPAP compliance | week 16
  the CPAP compliance is assessed in the two groups at week 16
Sleepiness | weeks 1 and 16
  Sleepiness is assessed with Epworth Sleepiness Scale at weeks 1 and 16 for the two groups
Physical Activity | week 1
  Daily Physical Activity is assessed with an accelerometer (Sensewear Armband, Bodymedia) at weeks 1 and 16 in the two groups. Daily expenditure, steps number, daily METs are assessed.
Quality of Life | week 16
  Quality of life is assessed with SF-12 questionnaire at weeks 1 and 16 in the two groups.
Cardiovascular risk SCORE | Week 1
  The cardiovascular risk SCORE is assessed at weeks 1 and 16 in the two groups.
Sleepiness | week 16
  Sleepiness is assessed with Epworth Sleepiness Scale at weeks 1 and 16 for the two groups
Physical Activity | week 16
  Daily Physical Activity is assessed with an accelerometer (Sensewear Armband, Bodymedia) at weeks 1 and 16 in the two groups. Daily expenditure, steps number, daily METs are assessed.
Quality of Life | week 1
  Quality of life is assessed with SF-12 questionnaire at weeks 1 and 16 in the two groups.
Cardiovascular risk SCORE | Week 16
  The cardiovascular risk SCORE is assessed at weeks 1 and 16 in the two groups.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Louis PEPIN, Prof, PhD, Principal Investigator — University Hospital, Grenoble
Locations (14):
- France (14):
  - Liberal Office, Boulogne-Billancourt
  - Clermont Tonerre military hospital, Brest
  - Liberal Office, Chambéry
  - Liberal Office, Grenoble
  - University Hospital, Grenoble
  - Liberal Office, Montigny-lès-Metz
  - Liberal Office, Nancy
  - Cornouaille Hospital, Quimper
  - Liberal Office, Saint Martin Les Boulogne
  - Montier Polyclinic, Saint-André-les-Vergers
  - Hospitalor Hospital, Saint-Avold
  - Liberal Office, Saint-Jean-de-Maurienne
  - Liberal Office, StIsmier
  - Liberal Office, Strasbourg

REFERENCES:
- [Derived] Mendelson M, Vivodtzev I, Tamisier R, Laplaud D, Dias-Domingos S, Baguet JP, Moreau L, Koltes C, Chavez L, De Lamberterie G, Herengt F, Levy P, Flore P, Pepin JL. CPAP treatment supported by telemedicine does not improve blood pressure in high cardiovascular risk OSA patients: a randomized, controlled trial. Sleep. 2014 Nov 1;37(11):1863-70. doi: 10.5665/sleep.4186. PMID 25364081
- [Derived] Mendelson M, Tamisier R, Laplaud D, Dias-Domingos S, Baguet JP, Moreau L, Koltes C, Chavez L, de Lamberterie G, Herengt F, Levy P, Flore P, Pepin JL. Low physical activity is a determinant for elevated blood pressure in high cardiovascular risk obstructive sleep apnea. Respir Care. 2014 Aug;59(8):1218-27. doi: 10.4187/respcare.02948. PMID 24282316